CLINICAL TRIAL: NCT07250542
Title: A Clinical Study on the Efficacy and Safety of Fasudil Hydrochloride Combined With Immunotherapy in the Treatment of Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: baotai Liang (Other)
Responsible Party: Sponsor-Investigator, baotai Liang, resident doctor, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024ZDSYLL151-P01
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The group treated with farsulide hydrochloride combined with immunotherapy (Experimental): This study is a single-arm clinical trial. Eligible patients will be included in the group receiving farsufilide hydrochloride combined with immunotherapy. After enrollment, in addition to the routine use of castration therapy, they will also receive farsufilide hydrochloride (10mg intravenous infusion) on days 1-5, and PD-1 monoclonal antibody (Tirapibep, 3mg/kg, intravenous infusion) on day 5. The treatment will be repeated every 21 days for a total of 4 times.
  Interventions: Drug: Fasudil hydrochloride combined with immunotherapy

INTERVENTIONS:
Drug: Fasudil hydrochloride combined with immunotherapy — This study is a single-arm clinical trial. Eligible patients will be included in the group receiving farsufilide hydrochloride combined with immunotherapy. After enrollment, in addition to the routine use of castration therapy, they will also receive farsufilide hydrochloride (10mg intravenous infusion) on days 1-5, and PD-1 monoclonal antibody (Tirapibep, 3mg/kg, intravenous infusion) on day 5. The treatment will be repeated every 21 days for a total of 4 times.

SUMMARY:
Carrying out clinical trials of salbutamol hydrochloride combined with immunotherapy and castration for the treatment of prostate cancer is of great significance. Firstly, it can verify the efficacy and safety of this combination in the treatment of prostate cancer, providing a scientific basis for its clinical application. Secondly, through clinical trials, the mechanism of action of salbutamol hydrochloride combined with immunotherapy can be further studied. Finally, this clinical trial can further expand the treatment strategies for prostate cancer.

DETAILED DESCRIPTION:
This study is a single-arm clinical trial. Eligible patients will be included in the group receiving farsufilide hydrochloride combined with immunotherapy. After enrollment, in addition to the routine androgen deprivation therapy, they will also receive farsufilide hydrochloride (10mg intravenous infusion) on days 1-5, and PD-1 monoclonal antibody (Tirapibep, 3mg/kg, intravenous infusion) on day 5. The treatment will be repeated every 21 days for a total of 4 times.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and < 85 years;
2. Patients who have failed at least one chemotherapy regimen containing docetaxel and one standard novel endocrine therapy;
3. Diagnosed with CRPC, defined as: after continuous castration therapy, the castration level of testosterone is < 50 ng/ml; disease progression within 12 weeks before enrollment: PSA levels increase consecutively for 3 times at intervals of 1 week, and serum PSA ≥ 2 ng/ml; evaluated as soft tissue progression according to RECIST criteria, or ≥ 2 new lesions on bone scan;
4. Imaging evidence indicates bone metastatic disease and/or measurable non-bone metastatic disease (lymph nodes or internal organs); Expected survival period ≥ 3 months; All patients voluntarily signed the informed consent form and were able to cooperate with treatment and follow-up;

Exclusion Criteria:

1. Severe cardiovascular and cerebrovascular diseases;
2. Abnormal liver function: Total bilirubin in blood is less than 1.5 times the upper limit of normal value, and the ratio of blood ALT to AST is less than 2 times the upper limit of normal value;
3. Abnormal kidney function: Serum creatinine is less than 1.5 mg/dl or the creatinine clearance rate is greater than or equal to 60 cc/min;
4. Those allergic to the used drugs;
5. Those with tumors in other parts;
6. Abnormal thyroid function: Blood FT4 and/or TT4 levels are higher or lower than the normal value (normal blood FT4 level is 9-25 pmol/L (0.7-1.9 ng/dl), normal blood TT4 level is 64-154 nmol/L (5-12 ug/dl));
7. Cortisol deficiency: Serum cortisol at 8 a.m. is less than 140 nmol/L (5 ug/dL).

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PSA level | About 4 months
  Before and after each cycle of treatment, blood samples were collected from the elbow vein on an empty stomach in the morning. The serum PSA level was detected using the enzyme-linked immunosorbent assay method.

SECONDARY OUTCOMES:
KPS scoring scale | About 4 months
  On the 6th day after medication administration, a quality of life assessment was conducted for the patient, referring to the KPS scoring scale. The score range is from 0 to 100, with 0 indicating death and 100 indicating normal, without any symptoms or signs. The assessment focused on the changes in the patient's quality of life, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, China